CLINICAL TRIAL: NCT05445154
Title: A Single-Arm, Multicenter, Open-Label, Dose- Escalating and Expanding,Phase I/II Study of SKLB1028 Combined With "7+3" Standard Chemotherapy in Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)
Brief Title: SKLB1028, Daunorubicin, and Cytarabine in Treating Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HA114-CSP-007
Record Dates: First submitted 2021-06-04; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-05

CONDITIONS: Newly Diagnosed Acute Myeloid Leukemia (AML)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SKLB1028 Dose Escalation (Experimental): Part1:Patients will receive a standard combination of chemotherapy drugs during remission induction therapy that includes cytarabine, daunorubicin, and the experimental drug SKLB1028.SKLB1028 capsules beginning at 100 mg bid.
  Part2: Once the appropriate therapeutic schedule has been established in Part 1, up to 20 subjects will be enrolled into an expansion cohort.
  Interventions: Drug: SKLB1028 Dose Escalation

INTERVENTIONS:
Drug: SKLB1028 Dose Escalation — Drug :SKLB1028 ;Drug: Cytarabine ;Drug: Daunorubicin

SUMMARY:
The purpose of this study is to describe the dose limiting toxicities (DLT) of SKLB1028 when combined with cytarabine/ daunorubicin remission induction in a 7+3 schedule. Safety and tolerability of SKLB1028 will also be evaluated. This study will also characterize the pharmacokinetics (PK) of SKLB1028 when given in combination with cytarabine/daunorubicin remission induction and high-dose cytarabine (HiDAC) consolidation therapy in newly diagnosed acute myeloid leukemia .

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a diagnosis of previously-untreated de novo acute myeloid leukemia (AML) > 20% blasts in the bone marrow according to WHO classification (2016) documented prior to enrollment.;
2. Age ≥ 18 and < 60 years;
3. Subjects who are positive for FLT3 mutations by central laboratory;
4. Subject has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;
5. Subject must meet the following criteria as indicated on the clinical laboratory tests;

   1. Serum aspartate aminotransf
   2. Total serum bilirubin ≤ 2.5 x institutional ULN
   3. Serum creatinine ≤ 3 x institutional ULN or an estimated glomerular filtration rate (eGFR) of > 30 ml/min
6. Subject is suitable for oral administration of study drug.

Exclusion Criteria:

1. Confirmed diagnosis of acute promyelocytic leukemia (M3 /APL), or BCR-ABL positive leukemia (ie, blast crisis of chronic myelogenous leukemia);
2. Diagnosis of active malignancy other than AML;
3. AML secondary to radiotherapy or chemotherapy for other tumors;
4. AML with central nervous system involvement;
5. Refractory hypokalemia or hypomagnesemia that is not easily corrected by symptomatic treatment and that occurs repeatedly in the past;
6. Current clinically significant graft-ve
7. Previous history of other malignancies.
8. Patients with clinically significant coagulation abnormalities, such as disseminated intravascular coagulation (DIC), hemophilia A, hemophilia B, and von Willebrand disease;
9. Major surgery of major organs has been performed before entering the study (for the definition of major surgery, refer to Grade 3 and 4 surgery specified in Management Measures for Clinical Application of Medical Technology, or the patient has not yet fully recovered from
10. Subject has received prior therapy for AML with the following exceptions: a. emergency leukapheresis; b. emergency treatment with hydroxyurea ;c. growth factor or cytokine support; d. steroid for anaphylaxis or transfusion reaction;

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLTs) | up to Day42
  A DLT is defined as any Grade ≥ 3 non-hematologic or extramedullary toxicity that occur during the DLT assessment period, and that is considered to be possibly, probably, or definitely related to onsolidation therapies including the study drugs.

SECONDARY OUTCOMES:
Pharmacokinetics profile of SKLB1028 | Days 8, 15, 18, and 21 for remission induction and Days 8, and 21 for consolidation and Days 1 for maintenance
  Observed trough concentration (Ctrough)
CR rate after the induction therapy | up to 3months
  CR is defined as a morphologically leukemia-free state at the post-baseline visit, having a neutrophil count of ≥ 1,000/mm^3 and platelet count of ≥ 100,000/mm^3, bone marrow blasts < 5%. There must be no evidence of Auer rods and no evidence of extramedullary leukemia.
Duration of remission | up to 24months
  Duration of remission included duration of composite complete remission (CRc), duration of complete remission (CR)/ complete remission with partial hematologic recovery (CRh), duration of CRh, duration of CR and duration of response (CRc + partial remission (PR).
Overall Survival | up to 60months
  OS was measured from the date of the first dose of treatment to the date of death from any cause or to the last date that the patient was known to be alive
Event-Free Survival | up to 24months
  EFS was defined as the time from randomization until treatment failure (Composite complete remission (CRc) or partial remission (PR) were not reached within 4 cycles), relapse (excluding relapse after PR), or death from any cause, whichever occurs first.
Leukemia-free survival | up to 24months
  The LFS was defined as the time from the date of first CR until the date of documented relapse (excluding relapse from PR) or death for participants who achieved CR (relapse date or death date - first CR disease assessment date + 1).
Rate of hematopoietic stem cell transplantation | up to 12months
  Transplantation rate is defined as the percentage of participants undergoing hematopoietic stem cell transplant (HSCT).

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, China